CLINICAL TRIAL: NCT06634810
Title: Comprehensive Patient-Centered Home-based Care Coaching for COPD Self-management
Acronym: SAMBA COPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Baystate Medical Center (Other); VNS Health (Unknown); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Alex D Federman, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY-23-00838; R01HL171695 (NIH); GCO-23-0270 (Other Grant/Funding Number: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2024-10-08; First posted 2024-10-10 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Home Based; Self Management; Pulmonary Rehabilitation; Coaching
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: This project will conduct a randomized controlled trial to evaluate a self-management support intervention for predominantly minoritized, low-income adults with COPD.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Research Coordinators conducting interviews, and all investigators will be blinded to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Selt-Management Support (SaMBA-COPD) (Experimental): Participants receiving SaMBA-COPD intervention by community health workers (CHW).
  Participants will receive comprehensive screening and targeted management of barriers to COPD control, incorporating home-based pulmonary rehabilitation, oral steroid and antibiotic prescribing for pre-emptive treatment of COPD exacerbations.
  Interventions: Behavioral: Self-Management Support
- Attention-Matched Support (Placebo Comparator): Participants will receive support by CHWs providing education using the COPD 1-2-3 booklet. Participants will receive similar visit frequencies but will not undergo barrier screening or targeted interventions.
  Interventions: Behavioral: COPD Education

INTERVENTIONS:
Behavioral: Self-Management Support — The intervention will be delivered by CHWs in person and supplemented with telephone or video encounters over 6 months. The intervention comprises six core elements: engagement, intake, self-management assessment, barrier screening, actions to address identified barriers, and follow-up/maintenance support.
  Other Names: SaMBA-COPD
  Arms: Selt-Management Support (SaMBA-COPD)
Behavioral: COPD Education — The attention control is where CHWs will provide COPD education using the COPD 1-2-3 booklet. The attention control will consist of 6 CHW visits (approximately 1 per month) with the patient and care giver in their home or via video conference, per patient preference.
  Arms: Attention-Matched Support

SUMMARY:
The Icahn School of Medicine at Mount Sinai will conduct a randomized controlled trial of a self-management support intervention for predominantly minoritized and low-income adults with chronic obstructive pulmonary disease (COPD). The trial will focus on comprehensive screening and targeted management of barriers to COPD control, incorporating home-based pulmonary rehabilitation and oral steroid and antibiotic prescribing for pre-emptive treatment of COPD exacerbations. The research team will compare this intervention with an attention control group to evaluate the effects on medication adherence, COPD symptoms, inhaler technique, physical activity and exercise capacity at 6 months, and at 12 months to examine sustainability of treatment effects. The research team will also examine hospitalizations and emergency department visits at 12 months. The study will recruit 300 participants from the Mount Sinai Health System in Manhattan, Queens, and Brooklyn, ensuring diverse representation. Health coaches from the VNS Health will deliver the intervention, guided by a detailed training manual. Weekly conference calls will address logistical and protocol-related issues.

DETAILED DESCRIPTION:
The Icahn School of Medicine at Mount Sinai is the lead and only site of recruitment for this project. Research study activities will be conducted at practices across the Mount Sinai Health System. The research team will identify a patient pool through the electronic health record. The research team will recruit 300 (150 per arm) participants from the Mount Sinai Health System in Manhattan, Queens, and Brooklyn in NYC. These practices provide care to a diverse population with considerable sociodemographic diversity (~40% Latino and ~30% Black, ~50% with household incomes <$1,350/month). Randomization will occur 1 month after the baseline interview (and after the devices are returned). Randomization will be in blocks of variable size (4 to 6) and stratified by Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria B or E. The study's main outcomes will be assessed at 6 months and sustainability of treatment effects at 12 months. The intervention will be delivered by community health workers (CHW)health coaches employed by VNS Health. The research team will follow a detailed intervention training manual and Manual of Operations to guide CHWs through the intervention. The CHWs will also attend a 90-minute monthly group meeting to discuss cases and hear presentations on topics of their choosing for skills and knowledge development. The research team will meet by conference call weekly to discuss logistical issues, refinement of protocol, and other issues pertaining to the study. The project manager will email any modifications to the IRB and research coordinator within one day of receiving approval. The project manager will also email a copy of the amendment approval letter. Mount Sinai will abide by IRB policies as serving site.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥40 years
* Chart-documented COPD with GOLD classifications B or E based on CAT score and number of exacerbations with or without hospitalization determined by electronic health record (EHR) review. GOLD class B and E patients are at increased risk of activity limiting symptoms and exacerbation and are more likely to benefit from the intensive SAMBA-COPD intervention.
* Prescribed a long-acting muscarinic agonist (LAMA), long-acting beta-adrenergic receptor agonist (LABA), an inhaled corticosteroid (ICS), or any combination of these since much of the intervention's focus is on medication adherence.
* English or Spanish speaking

Exclusion Criteria:

* EHR documented dementia, as the research teams focus is on patients with capacity to independently perform self-care tasks.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
COPD Assessment Test (CAT) Score | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  The COPD Assessment Test (CAT) is a validated measure of the impact of COPD on a person's life. COPD symptoms will be measured by self-report using the CAT. Full range from 0-40, with higher scores indicating a more severe impact of COPD on a patient's life.
Number of participants who adhere to ≥ 80% of prescribed actuations | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  Adherence will be measured by the number of participants who adhere to ≥ 80% of prescribed actuations (doses).

SECONDARY OUTCOMES:
Inhaler Technique | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  Participants will be observed performing an inhalation from their COPD controller medication. Participant inhaler technique will be scored using a validated checklist. Higher score indicates better health outcomes.
  For metered dose and dry powdered inhalers, 0-7
  For Ellipta devices, 0-9
  For Respimat devices, 0-12
Number of steps counted on Actigraph | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  Physical activity will be measured by total number of steps counted on triaxial accelerometer (Actigraph).
Quality of life measured using the Clinical COPD Questionnaire (CCQ) | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  The CCQ is a 10-item questionnaire scored from 0 to 6 for each item (0 being never and 6 being all the time, with higher scores representing worse quality of life). The total score is 0-60.
Number of participants with hospitalizations | at Baseline and at 12 months
  Number of participants with hospitalizations for COPD-related events obtained from the Statewide Planning and Research Cooperative System (SPARCS).
Number of participants with emergency department (ED) visits | at Baseline and at 12 months
  Number of participants with ED visits obtained from the Statewide Planning and Research Cooperative System (SPARCS).
Six Minute Walk Test (6MWT) to measure Exercise Capacity | at baseline, end of treatment period (each treatment period are 90-minute monthly treatments over 6 months), and 6 months after end of treatment period
  The 6MWT measures the total the distance walked by the participant over 6 minutes on a closed track.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Federman, MD, MPH, Principal Investigator — Ichan School of Medicine at Mount Sinai, The Mount Sinai Hospital
Locations (1):
- Ichan School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Study data will be made available to other users after publication of the study's main results (primary analyses of Aims 1-3). Once made available, no time limit will be placed on accessibility of the study data.
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (Link to be included in the URL field below).

REFERENCES:
- [Derived] Agrawal N, Case M, Lindenauer PK, McDermott D, Diaz KM, Utkin JO, Wisnivesky J, Federman A. Protocol for a randomized trial of self-management support for people with chronic obstructive pulmonary disease using lay health coaches. Contemp Clin Trials. 2025 Nov;158:108095. doi: 10.1016/j.cct.2025.108095. Epub 2025 Sep 22. PMID 40992542